CLINICAL TRIAL: NCT04898309
Title: A Placebo-controlled Randomized Trial to Evaluate the Efficacy and Safety of GNR-038 in Comparison With Berinert® for Acute Attacks Relief in Patients With Hereditary Angioedema
Brief Title: Efficacy and Safety of GNR-038 vs Berinert® in Patients With Hereditary Angioedema
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Company pipeline revision
Sponsor: AO GENERIUM (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIR-HAE-II-III; #210, April 16, 2 (Other: Ministry of Health of Russian Federation)
Record Dates: First submitted 2021-05-18; First posted 2021-05-24 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Hereditary Angioedema
Keywords: Hereditary angioedema; Swelling; GNR-038; C1-inhibitor; Mutation; SERPING1 gene; HAE; Genetic disease; C1-INH deficiency; Hypersensitivity; Immune System Diseases; Genetic Diseases, Inborn; Immunologic Factors; Physiological Effects of Drugs; Complement Inactivating Agents; Immunosuppressive Agents; Angioedema; Angioedemas, Hereditary; Complement C1 Inhibitor Protein; Complement C1 Inactivator Proteins
MeSH Terms: conditions — Angioedemas, Hereditary; Genetic Diseases, Inborn; Hypersensitivity; Immune System Diseases; Angioedema | interventions — Complement C1 Inhibitor Protein

STUDY DESIGN:
Intervention Model Description: Two-stage study. In the first stage - 4 groups are presented. At the second stage - 2 study groups 200 HAE attacks to be randomized in 50 patients
Who Masked: Participant, Investigator
Masking Description: At the first stage - the study will be blinded, at the second stage - open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Study stage 1: GNR-038, 50 МЕ/ kg (Experimental): Recombinant C1 esterase inhibitor
  Interventions: Drug: GNR-038, 50 МЕ/ kg
- Study stage 1: GNR-038, 100 МЕ/ kg (Experimental): Recombinant C1 esterase inhibitor
  Interventions: Drug: GNR-038, 100 МЕ/ kg
- Study stage 1: Berinert®, 20 МЕ/ kg (Experimental): Human C1 esterase inhibitor
  Interventions: Drug: Berinert®, 20 МЕ/ kg
- Study stage 1: Placebo (Experimental): Placebo
  Interventions: Drug: Placebo
- Study stage 2: GNR-038 in selected dose (Experimental): Recombinant C1 esterase inhibitor
  Interventions: Drug: GNR-038. The dose will be selected according to results of stage 1 clinical trial.
- Study stage 2: Berinert®, 20 МЕ/ kg (Experimental): Human C1 esterase inhibitor
  Interventions: Drug: Berinert®, 20 МЕ/ kg

INTERVENTIONS:
Drug: GNR-038, 50 МЕ/ kg — A single intravenous infusion of GNR-038, 50 МЕ/ kg less than 5 hours after the onset of edema.
  Other Names: Recombinant C1 esterase inhibitor, 50 МЕ/ kg
  Arms: Study stage 1: GNR-038, 50 МЕ/ kg
Drug: GNR-038, 100 МЕ/ kg — A single intravenous infusion of GNR-038, 100 МЕ/ kg less than 5 hours after the onset of edema.
  Other Names: Recombinant C1 esterase inhibitor, 100 МЕ/ kg
  Arms: Study stage 1: GNR-038, 100 МЕ/ kg
Drug: Berinert®, 20 МЕ/ kg — A single intravenous infusion of Berinert®, 20 МЕ/ kg less than 5 hours after the onset of edema.
  Other Names: Human C1 esterase inhibitor
  Arms: Study stage 1: Berinert®, 20 МЕ/ kg
Drug: Placebo — A single intravenous infusion of Placebo less than 5 hours after the onset of edema.
  Arms: Study stage 1: Placebo
Drug: GNR-038. The dose will be selected according to results of stage 1 clinical trial. — A single intravenous infusion of GNR-038 less than 5 hours after the onset of edema.
  Other Names: Recombinant C1 esterase inhibitor.
  Arms: Study stage 2: GNR-038 in selected dose
Drug: Berinert®, 20 МЕ/ kg — A single intravenous infusion of Berinert®, 20 МЕ/ kg less than 5 hours after the onset of edema.
  Other Names: Human C1 esterase inhibitor
  Arms: Study stage 2: Berinert®, 20 МЕ/ kg

SUMMARY:
It is a placebo-controlled randomized trial to evaluate the efficacy and safety of GNR-038 in comparison with Berinert® in patients with hereditary angioedema

DETAILED DESCRIPTION:
Hereditary angioedema is a rare, potentially life-threatening genetically determined disease associated with a deficiency or impairment of the functional activity of the C1-esterase inhibitor (C1-inhibitor). The main clinical manifestation of hereditary angioedema is recurrent subcutaneous or submucosal swelling of various localization. Most often, the development of the disease is based on a mutation in the SERPING1 gene. The prevalence of the disease in the world ranges from 1:10 000 to 1:150 000. GNR-038 is a recombinant C1 inhibitor (rhC1INH), which is a complete structural and functional analog of the plasma C1 inhibitor. Phase I study results showed convincing safety and tolerability evidence of GNR-038.

ELIGIBILITY:
Inclusion Criteria

1. Men and women 18 years and older at the time of signing the Informed Consent Form.
2. Availability of written informed consent signed by the patient prior to the start of any procedures related to the study.
3. Confirmed diagnosis of HAE:

   * C4 level <50% of the lower limit of the range of normal laboratory values and one of the points below:
   * the C1INH level <50% of the lower limit of the range of normal laboratory values, OR
   * the level of C1INH within normal values, while the level of functional activity of C1INH is below 50% of the lower limit of the range of normal values.
4. Localization of the edema in the abdominal cavity, in the face area (lips, eyelids, subcutaneous tissue), limbs, trunk or in the area of the external genitals in the anamnesis.
5. ≥4 HAE attacks requiring treatment or causing significant functional impairment for 2 consecutive months in the 3-month period prior to Screening, properly documented in the medical records.
6. Patient's consent to adhere to reliable methods of contraception.

Exclusion Criteria

1. Deviation of the C1q level below the normal limit.
2. B-cell lymphoproliferative diseases in the anamnesis or at the time of inclusion in clinical trial.
3. The presence of anti-C1INH autoantibodies.
4. Allergic reactions to the components of C1INH drugs or other blood components.
5. Glomerular filtration rate ≤59 ml/min/1.73 m2, calculated by the formula CKD-EPI Creatinine Equation (2009) (see Appendix).
6. The concentration of peripheral blood leukocytes >20*109/L.
7. Drug addiction, solvent abuse, alcoholism in the anamnesis or at the time of inclusion.
8. Participation in clinical trials of C1-esterase inhibitor drugs, blood transfusion and its components during the last 90 days prior to screening.
9. Participation in clinical trials of any other investigational drugs within the last 30 (thirty) days prior to screening.
10. Positive laboratory results for HIV and hepatitis B and C.
11. Pregnancy and lactation.
12. Diseases and conditions associated with thrombosis (myocardial infarction, transient ischemic attacks, deep and superficial vein thrombosis, and pulmonary embolism) less than 6 months before the start of the screening period, as well as an increased risk of arterial or venous thrombosis according to the study doctor's opinion.
13. Concomitant diseases and conditions that according to the study doctor's opinion put the patient's safety at risk when participating in the study, or that will affect the analysis of safety data if this disease/condition worsens during the study, including:

    * Mental illness;
    * Diseases of the immune and endocrine system that are not controlled by drug therapy (including decompensated diabetes mellitus and thyroid diseases);
    * Hematological diseases requiring chemotherapy;
    * Cancer or cancer in the past medical history, with the exception of cured basal cell carcinoma;
    * Decompensated liver diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Time to symptoms relief onset of acute HAE attack within 24 hours after the end of the drug administration. | 24 hours
  A persistent decrease in the intensity of symptoms by 20 mm from the initial level on the visual analogue scale (VAS) will be regarded as a relief of symptoms of HAE. 0 mm is the absence of symptoms, 100 mm is the maximum possible intensity of symptoms

SECONDARY OUTCOMES:
Time to complete resolution of the symptoms of an acute HAE attack within 24 hours after the end of the study drug administration. | 24 hours
  Persistent absence of symptoms - 0 (zero) mm on the visual analogue scale (VAS). 0 mm is the absence of symptoms, 100 mm is the maximum possible intensity of symptoms
Time to minimum manifestation onset of acute HAE attack symptoms after the completion of study drug administration. | 24 hours
  Persistent reduction in the intensity of symptoms below 20 (twenty) mm on the visual analogue scale(VAS). 0 mm is the absence of symptoms, 100 mm is the maximum possible intensity of symptoms
The proportion of HAE exacerbation episodes that achieved symptom relief after 1 hour and 4 (four) hours after the end of study drug administration. | 1 hour; 4 hours.
The rate of attacks with HAE current localization relapse or with the occurrence of a new acute attack of a different localization within 24 (twenty-four) hours after the study drug administration. | 24 hours
The rate of attacks that required additional administration of emergency drugs (human C1-esterase inhibitor or icatibant). | 24 hours
The rate of attacks that did not respond therapeutically to the study drug administration | 4 hours; 24 hours
  the lack of relief of HAE symptoms within 4 (four) hours after administration of the drug, the occurrence of a relapse of HAE of the current localization or the occurrence of a new acute attack of another localization within 24 (twenty-four) hours after drug administration, the need to use drugs that can weaken the symptoms of HAE (see drugs that are not recommended to treatment), within 24 (twenty-four) hours after drug administration.
The intensity of acute HAE attack symptoms within 24 (twenty-four) hours after study drug administration. | 24 hours
  HAE intensity wiil be measured by visual analogue scale (VAS). 0 mm is the absence of symptoms, 100 mm is the maximum possible intensity of symptoms
Frequency of adverse events. | 14 days
Frequency of anti-drug antibody formation. | 7 and 14 days
The level of anti-drug antibodies neutralizing activity. | 7 and 14 days
  Laboratory measurement of antidrug antibody with neutralixing activity.

CONTACTS AND LOCATIONS:
Overall Officials: Oksana A. Markova, MD, Study Chair — AO GENERIUM
Locations (5):
- Russia (5):
  - National Research Center - Institute of Immunology Federal Medical-Biological Agency of Russia, Moscow
  - Moscow City Clinical Hospital 52, Moscow
  - Federal State Budgetary Scientific Institution Research Institute of Fundamental and Clinical Immunology, Moscow
  - Rostov State Medical University, Rostov-on-Don
  - LLC "Scientific Medical Center of General Therapy and Pharmacology", Stavropol

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical trial registry, Ministry of Health of Russian Federation — https://grls.rosminzdrav.ru/CIPermissionMini.aspx?CIStatementGUID=fdafdfaf-8475-4d3e-810a-e18d4fc64236&CIPermGUID=AEE75E93-3F3E-4A76-8EB1-B57F8C5A48C0
- See also: Clinical trial registry — https://clinline.ru/reestr-klinicheskih-issledovanij/210-16.04.2021.html